CLINICAL TRIAL: NCT01666236
Title: Triple Treatment for Detachment of Retinal Pigment Epithelium Secondary to Polypoidal Choroidal Vasculopathy.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of resources
Sponsor: Federal University of São Paulo (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Dr. Pedro Paulo de Oliveira Bonomo, phD, Federal University of São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBPD952ABR01T
Record Dates: First submitted 2012-08-08; First posted 2012-08-16 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Choroidal Neovascularization; Retinal Pigment Epithelial Detachment
Keywords: Age-Related Macular Degeneration; Pigment Epithelial Detachment; Polypoidal Choroidal Vasculopathy
MeSH Terms: conditions — Choroidal Neovascularization; Retinal Detachment; Macular Degeneration; Polypoidal Choroidal Vasculopathy | interventions — Verteporfin; Ranibizumab; Triamcinolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Triple Therapy (Other): The treatment (single group) will be treated with reduced-fluence Photodynamic Therapy (Visudyne -Verteporfin infused over 10 minutes at a dose of 6mg/m2 and following by activating light [wavelength of 689 nm] applied 15 minutes after the start of infusion with a light dose of either 25 J/cm2 for 83 seconds), followed by an Intra-vitreous triamcinolone (4mg/0.1ml) on the same day.
  After 10 days, patients will be subjected to an injection of Intra-vitreous ranibizumab (0.5 mg/0.05 ml). After this first injection, Intra-vitreous ranibizumab will be repeated twice, on a monthly basis, for a total of three injections
  Interventions: Other: Triple Therapy

INTERVENTIONS:
Other: Triple Therapy — The treatment (single group) will be treated with reduced-fluence Photodynamic Therapy (Visudyne -Verteporfin infused over 10 minutes at a dose of 6mg/m2 and following by activating light [wavelength of 689 nm] applied 15 minutes after the start of infusion with a light dose of either 25 J/cm2 for 83 seconds), followed by an Intra-vitreous triamcinolone (4mg/0.1ml) on the same day.
  After 10 days, patients will be subjected to an injection of Intra-vitreous ranibizumab (0.5 mg/0.05 ml). After this first injection, Intra-vitreous ranibizumab will be repeated twice, on a monthly basis, for a total of three injections
  Other Names: Verteporfin; Ranibizumab; Triamcinolone

SUMMARY:
Study the effectiveness of the treatment detachment of retinal pigment epithelium secondary to polypoidal choroidal vasculopathy. Efficacy will be assessed by regression of polyp area after twelve months, compared to baseline. Treatment under study is a triple therapy with: 1) reduced-fluence photodynamic therapy (PDT), 2) intravitreal (IVT) triamcinolone and, 3) IVT ranibizumab, for the treatment of detachment of the retinal pigment epithelium (PED) secondary to Polypoidal Choroidal Vasculopathy (PCV).

ELIGIBILITY:
Inclusion Criteria:

* Patients with PCV associated with PED near the polypoidal lesion recently diagnosed, documented by FA, ICGA and OCT.
* Visual acuity between 20/40 and 20/400.
* Patients older than 50 years (both genders).
* Women must be postmenopausal for at least 12 months or surgically sterile.
* No previous treatment in the study eye.
* Accept and sign the informed consent.
* No condition that prevents the monitoring of the patient for one year.
* Transparent ocular media and adequate pupillary dilation to allow good images of the fundus.

Exclusion Criteria:

* Blepharitis or external eye infection.
* Allergy to ranibizumab, verteporfin, triamcinolone, fluorescein or indocyanine green.
* Patients unable to provide informed consent.
* Concomitant ocular disease that impairs visual acuity.
* Any intraocular condition (such as cataract or Proliferative Diabetic Retinopathy) in the study eye, in the opinion of the investigator, could require surgery or medication during the follow-up (1 year).
* Active intraocular inflammation.
* Patients with Glaucoma and with ocular hypertension (IOP > 25mmHg).
* Premenopausal women. Pregnancy or lactation.
* Effective treatment for active systemic infection or history of recurrent infection.
* Evidence of concomitant disease (cardiovascular, neurological, pulmonary, renal, hepatic, endocrine or gastrointestinal) uncontrolled.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Auxiliary Exams - Optical Coherency Tomography (OCT) | 12 months after first procedure
  Optical Coherency Tomography (OCT): To Assess the Retinal Thickness using the ETDRS thickness profile and to evaluate the regression of the pigment epithelium detachment.
  The Auxiliary exams are done at the Baseline, 10 days after the procedure and every 30 days until the end of the study.
Auxiliary Exams - Indocyanine green angiography (ICGA) | 12 months after first procedure
  Indocyanine green angiography (ICGA): To Evaluate the polyp lesions regression
  The Auxiliary exams are done at the Baseline, 10 days after the procedure and every 30 days until the end of the study.
Auxiliary Exams - Fluorescein Angiography (FA) | 12 months after first procedure
  Fluorescein Angiography (FA): To Evaluate subretinal neovascularization
  The Auxiliary exams are done at the Baseline, 10 days after the procedure and every 30 days until the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Paulo O Bonomo, phD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Universidade Federal de São Paulo - Escola Paulista de Medicina, São Paulo, São Paulo, Brazil

REFERENCES:
- [Result] 1. Bessho H, Honda S, Imai H, Negi B. Natural Course and Funduscopic Findings of Polypoidal Choroidal Vasculopathy in a Japanese Population Over 1 Year of Follow-up. Retina 2011; X: 1-5. 2. Uyama M, Wada M, Nagai Y, Matsubara T, Matsunaga H, Fukushima I, Takahashi K, Matsumura AM. Polypoidal Choroidal Vasculopathy: Natural History. Am J Ophthalmol 2002 May;133(5):639-648. 3. Ruamviboonsuk P, Tadarati M, Vanichvaranont S, Hanutsaha P, Pokawattana N. Photodynamic therapy combined with ranibizumab for polypoidal choroidal vasculopathy: results of a 1-year preliminary study. Br J Ophthalmol 2010;94:1045-1051. 4. Hikichi T, Ohtsuka H, Higuchi M, Matsushita T, Ariga H, Kosaka S, Matsushita R, Takami K. Improvement of Angiographic Findings of Polypoidal Choroidal Vasculopathy After Intravitreal Injection of Ranibizumab Monthly for 3 Months. Am J Ophthalmol 2010 Nov;150(5):674-682. 5. Kovacs KD, Quirk MT, Kinoshita T, Gautam S, Ceron OM, Murtha TJ, Arroyo JG. A retrospective analysis of triple combination therapy with intravitreal bevacizumab, posterior sub-tenon's triamcinolone acetonide, and low-fluence verteporfin photodynamic therapy in patients with neovascular age-related macular degeneration. Retina 2011 Mar;31(3):446-52. 6. Becerra EM, Morescalchi F, Gandolfo F, Danzi P, Nascimbeni G, Arcidiacono B, Semeraro F. Clinical evidence of intravitreal triamcinolone acetonide in the management of age-related macular degeneration. Curr Drug Targets. 2011 Feb;12(2):149-72. 7. Hajouli N, Hiesch A, Quintyn JC. Triple therapy for the treatment of choroidal neovascularization with pigment epithelium detachment in age-related macular degeneration. J Fr Ophtalmol. 2010 Sep;33(7):487-92. 8. Tao Y, Jonas JB. Intravitreal bevacizumab combined with intravitreal triamcinolone for therapy-resistant exudative age-related macular degeneration. J Ocul Pharmacol Ther. 2010 Apr;26(2):207-12.